CLINICAL TRIAL: NCT00332449
Title: Does Early Breast Feeding Prevents Neonatal Hypoglycemia in High Risk Newborns
Brief Title: Early Breast Feeding and Glucose Levels in High Risk Newborns
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Ayala Maayan, Sheba Medical Center
Other Study IDs: SHEBA-06-4112-AM-CTIL
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Neonatal Hypoglycemia
Keywords: early breast feeding; hypoglycemia; newborn
MeSH Terms: conditions — Breast Feeding; Hypoglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Early breast feeding has shown to be important to mother-infant bonding and is associated with longer duration of breast feeding. However, little data is available regarding its contribution to glucose levels in the newborn infants. Newborns that are at risk to develop hypoglycemia may benefit from early breast feeding if this appears to prevent post-partum hypoglycemia.

DETAILED DESCRIPTION:
Mothers will be encouraged to breast feed early after delivery (at the delivery room). Data of high risk babies for developing post partum hypoglycemia (Infants of diabetic mothers, infants of hypertensive mothers, infants with birth weight more than 4 Kg or less than 2.5 Kg and infants with meconium stained amniotic fluid)will be recorded including maternal breast feeding times and quality of feeding. Glucose levels shall be routinely monitored and recorded at the neonatal department. A comparison of all data will be made between those newborns that breast feed after labor and those who were not.

ELIGIBILITY:
Inclusion Criteria:

* Newborns to diabetic mothers
* Newborns to hypertensive mothers
* Newborns with birth weight greater than 4 Kg or less than 2.5 Kg
* Newborns with meconium stained amniotic fluid

Exclusion Criteria:

* Newborns with major congenital malformation
* Preterm babies
* Newborns with post-birth distress

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary clinic clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-06 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
normal neonatal glucose levels | 2 days

SECONDARY OUTCOMES:
Hypoglycemia prevention | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Ayala Maayan-Metzger, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center - Neonatal Department, Ramat Gan, Tel-Hashomer, Israel